CLINICAL TRIAL: NCT00266682
Title: Clinical Investigation of the SelectSecure Pacing Lead
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 600
Record Dates: First submitted 2005-12-16; First posted 2005-12-19 (Estimated); Last update posted 2006-10-13 (Estimated); Status verified 2006-10

CONDITIONS: Bradycardia
Keywords: Bradycardia
MeSH Terms: conditions — Bradycardia

INTERVENTIONS:
Device: Pacing Lead

SUMMARY:
People who have a slow heart beat, or whose heart does not beat on its own, may be in need of an electronic device called a pacemaker. A pacemaker is implanted surgically just under the skin in the upper chest area. This device helps the heart beat at a regular rhythm by sending electrical signals (pacing) directly to the heart tissue through flexible wires called leads. The purpose of this study is to demonstrate that the SelectSecure (Model 3830) lead is safe and effective for both sensing the heart's natural rhythm and pacing the heart when it does not beat on its own. This lead will be studied in both the right atrium and right ventricle. A previously market approved Medtronic lead model will serve as a comparison to prove the safety and effectiveness of the SelectSecure Model.

ELIGIBILITY:
Inclusion Criteria:

Subjects who are in need of a pacemaker that paces in both the right atrium and ventricle.

Exclusion Criteria:

Subjects who are in need of an implantable cardioverter defibrillator (ICD).

Subjects who have a mechanical or diseased tricuspid valve (a structure in the heart, located between the right atrium and right ventricle, which allows blood to flow from the atrium to the ventricle).

Steroid contraindication

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 365
Dates: Start 2002-08; Study Completion 2005-08

PRIMARY OUTCOMES:
3-month safety (complications and all lead-related adverse events) and efficacy ( pacing and sensing) objectives

SECONDARY OUTCOMES:
Lead and catheter handling characteristics, and lead impedance

CONTACTS AND LOCATIONS:
Locations (31):
- United States (26):
  - Anchorage, Alaska
  - Peoria, Arizona
  - Long Beach, California
  - Santa Rosa, California
  - Fort Lauderdale, Florida
  - Evanston, Illinois
  - Indianapolis, Indiana
  - Des Moines, Iowa
  - Iowa City, Iowa
  - Kansas City, Kansas
  - Boston, Massachusetts
  - Detroit, Michigan
  - Robbinsdale, Minnesota
  - Saint Paul, Minnesota
  - Kansas City, Missouri
  - Springfield, Missouri
  - Livingston, New Jersey
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Lancaster, Pennsylvania
  - Sayre, Pennsylvania
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Temple, Texas
  - Richmond, Virginia
- Melbourne, Australia
- Canada (4):
  - Kingston
  - London
  - Ottawa
  - Sainte-Foy